CLINICAL TRIAL: NCT06288412
Title: Pharmacodynamic Properties of Insulin Icodec During Exercise and Prolonged Fasting in Participants With Type 2 Diabetes
Brief Title: A Study to Test How a New Long-acting Insulin Works in the Body of Patients With Type 2 Diabetes During Exercise and Prolonged Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-7615; U1111-1285-1665 (Other: World Health Organization (WHO)); 2023-505012-38 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Insulin icodec (Experimental): Participants will receive subcutaneous (s.c.) injections of insulin degludec once daily in the run-in period and insulin icodec once weekly in the treatment period.
  Interventions: Drug: Insulin icodec; Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive insulin icodec subcutaneous (s.c.) once weekly.
Drug: Insulin degludec — Participants will receive insulin degludec s.c. once daily.

SUMMARY:
The study will investigate the safety of once weekly insulin icodec subcutaenously (s.c.) during and after exercise and prolonged fasting in patients with type 2 diabetes (T2D). Participants will first receive insulin decludec (Tresiba®, a long-acting insulin taken once daily) for atleast one week. Afterwards participants will receive insulin icodec that will be administered once weekly at the study site (for a minimum of 7 weeks and maximum of 14 weeks). Insulin icodec is a novel long-acting insulin analogue for once-weekly administration for the treatment of type 2 diabetes. The study will last for about 16-30 weeks. Participant must not participate if participant have suspected hypersensitivity reactions to the study products or cardiovascular diseases within the last 180 days. Female participant cannot take part if she is pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female.
* Age 18-75 years (both inclusive) at the time of signing the informed consent.
* Body mass index between 18.0 and 38.0 kilogram per meter^2 (kg/m^2) (both inclusive).
* Glycated hemoglobin (HbA1c) less than or equal to (<=) 9 percent (75 millimoles per mole [mmol/mol]) at screening.
* Treated with basal insulin with or without any of the following anti-diabetic drugs/regimens with stable doses >= 90 days prior to the day of screening:

  * Metformin,
  * Dipeptidyl peptidase 4 (DPP-4) inhibitors,
  * Sodium-Glucose Transport Protein 2 (SGLT2) inhibitors
* Oral combination products (for the allowed individual oral antidiabetic drugs), Injectable and oral glucagon-like peptide 1 (GLP-1) Receptor Agonists.
* Physically active >= 300 metabolic equivalent of task (MET) minutes/week as determined by an International Physical Activity Questionnaire (IPAQ) at screening.
* Mass-specific oxygen volume (VO2) peak greater than (>) 25 milliliters per kilogram per minute (mL/kg/min) as determined by cardiopulmonary testing (CPX) test at screening.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method.
* Presence or history of cardiovascular disease including stable and unstable angina pectoris, myocardial infarction, transient ischaemic attack, stroke, cardiac decompensation, clinically significant arrhythmias or clinically significant conduction disorders within 180 days prior to the day of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Time below range, glucose less than (<) 3.0 millimoles per liter (mmol/L) (54 milligrams per deciliter [mg/dL]) within 24 hours after start of exercise (TBR3.0mmol/L,exe) | 0-24 hours after start of exercise at Day 38
  Measured in percentage of readings.

SECONDARY OUTCOMES:
Time below range, glucose <3.9 mmol/L (70 mg/dL) within 24 hours after start of exercise (TBR3.9mmol/L,exe) | 0-24 hours after start of exercise at Day 38
  Measured in percentage of readings.
Time in range, glucose 3.9-10.0 mmol/L (70-180 mg/dL) within 24 hours after start of exercise (TIR3.9-10.0mmol/L,exe) | 0-24 hours after start of exercise at Day 38
  Measured in percentage of readings.
Time above range, glucose >10 mmol/L (180 mg/dL) within 24 hours after start of exercise (TAR10.0mmol/L,exe) | 0-24 hours after start of exercise at Day 38
  Measured in percentage of readings.
Number of clinically significant hypoglycaemic episodes during exercise (Hypoexe) | 0-40 minutes after start of exercise at Day 38
  Measured as number of episodes.
Amount of carbohydrate intake during exercise (CHOexe) | 0-40 minutes after start of exercise at Day 38
  Measured in gram (g).
Amount of carbohydrate intake from end of standardised lunch meal until start of exercise (CHOpre-exe) | 0-90 minutes before start of exercise at Day 38
  Measured in g.
Amount of carbohydrate intake after stop of exercise until start of standardised dinner meal (CHOpost-exe) | 0-140 minutes after start of exercise at Day 38
  Measured in g.
Number of hypoglycaemic within 24 hours after start of exercise (Hypo24h,exe) | 0-24 hours after start of exercise at Day 38
  Measured as number of episodes.
Number of hypoglycaemic episodes for 24 hours in reference week (43 to 67 hours after dosing) (Hypo24h,ref) | 43-67 hours after dosing at Day 29
  Measured as number of episodes.
Time below range, glucose <3.0 mmol/L (54 mg/dL) within 18 hours after start of fasting (TBR3.0mmol/L,fast) | 0-18 hours after start of fasting at Day 44
  Measured in percentage of readings.
Time below range, glucose <3.9 mmol/L (70 mg/dL) within 18 hours after start of fasting (TBR3.9mmol/L,fast) | 0-18 hours after start of fasting at Day 44
  Measured in percentage of readings.
Time in range, glucose 3.9-10 mmol/L (70-180 mg/dL) within 18 hours after start of fasting (TIR3.9-10.0mmol/L,fast) | 0-18 hours after start of fasting at Day 44
  Measured in percentage of readings.
Time above range, glucose >10 mmol/L (180 mg/dL) within 18 hours after start of fasting (TAR10.0mmol/L,fast) | 0-18 hours after start of fasting at Day 44
  Measured in percentage of readings.
Number of clinically significant hypoglycaemic episodes during fasting (Hypofast) | 0-18 hours after start of fasting at Day 44
  Measured as number of episodes.
Amount of carbohydrate administered intravenously during fasting (CHOfast) | 0-18 hours after start of fasting at Day 44
  Measured in g.
Number of hypoglycaemic episodes within 18 hours after start of fasting (Hypo18h,fast) | 0-18 hours after start of fasting at Day 44
  Measured as number of episodes.
Number of hypoglycaemic episodes for 18 hours in reference week (26 to 44 hours after dosing) (Hypo18h,ref) | 26-44 hours after dosing at Day 29
  Measured as number of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com